CLINICAL TRIAL: NCT04969211
Title: An Open-Label, Two-Period, Randomized, Single Oral Dose, Crossover Study to Evaluate the Bioequivalence of VHX-896 Tablets Relative to Iloperidone Tablets in Healthy Volunteers
Brief Title: Bioequivalence Study Between VHX-896 Tablets and Iloperidone Tablets in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VP-VHX-896-1101
Record Dates: First submitted 2021-07-09; First posted 2021-07-20 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Healthy
Keywords: Iloperidone; VHX-896; Bioequivalence
MeSH Terms: interventions — iloperidone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence A: VHX-896 then iloperidone (Experimental)
  Interventions: Drug: VHX-896 and iloperidone
- Sequence B: Iloperidone then VHX-896 (Experimental)
  Interventions: Drug: Iloperidone and VHX-896

INTERVENTIONS:
Drug: VHX-896 and iloperidone — oral tablet
  Arms: Sequence A: VHX-896 then iloperidone
Drug: Iloperidone and VHX-896 — oral tablet
  Arms: Sequence B: Iloperidone then VHX-896

SUMMARY:
This is a single center, two-period, randomized study to evaluate the Bioequivalence of VHX-896 Tablets Relative to Iloperidone Tablets in Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female participants between 18 to 55 years (inclusive).
* Have a Body Mass Index (BMI) of > 18.0 and < 30.0 kg/m2; (BMI = weight (kg)/ [height (m)]2).
* Good health as determined by no clinically significant deviations from normal in medical history, clinical laboratory determination, ECGs, and physical examinations conducted during the screening visit.
* Participants with no clinically significant medical, psychiatric or sleep disorders as determined by the PI.

Exclusion Criteria:

* Participants with history of drug or alcohol abuse within the 12 months prior to dosing or evidence of such abuse as indicated by the laboratory assays conducted during the screening or baseline evaluations.
* Participants who suffered from significant physical illness (required hospitalization) in the 4-week period preceding baseline will be excluded.
* Pregnant or nursing (lactating) women.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2021-10-13 (Actual)

PRIMARY OUTCOMES:
Bioequivalence between VHX-896 tablets relative to iloperidone tablets | 96 hours
  as measured by plasma concentrations
Assessment of Safety and Tolerability of a single dose of VHX-896 | 17 days
  As measured by the incidence of adverse events and clinically significant changes in laboratory values, ECG parameters, and vital signs

CONTACTS AND LOCATIONS:
Locations (1):
- Vanda Investigational Site, Springfield, Missouri, United States

IPD SHARING:
Plan to Share IPD: No